CLINICAL TRIAL: NCT00807937
Title: A Multi-Center, Randomized, Placebo-Controlled, Double-Blind, Parallel Group, Phase II Study of 2 Oral Dose Groups of AZD7325, With a Lorazepam Arm, in Subjects With Generalized Anxiety Disorder (GAD)
Brief Title: Proof of Concept in Patients With Generalized Anxiety Disorder (GAD)AZD7325
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Mark A. Smith, MD PhD, Medical Science Director, Emerging Psychiatry, AstraZeneca Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D1140C00014
Record Dates: First submitted 2008-12-12; First posted 2008-12-15 (Estimated); Results first posted 2010-10-08 (Estimated); Last update posted 2010-10-08 (Estimated); Status verified 2010-09

CONDITIONS: Anxiety Disorders
Keywords: Generalized Anxiety Disorder; GAD; Anxiety
MeSH Terms: conditions — Anxiety Disorders; Generalized Anxiety Disorder | interventions — 4-amino-8-(2-fluoro-6-methoxy-phenyl)-N-propylcinnoline-3-carboxamide; Lorazepam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- A (Experimental): AZD7325 5mg twice daily
  Interventions: Drug: AZD7325
- B (Experimental): AZD7325 15mg twice daily
  Interventions: Drug: AZD7325
- C (Active Comparator): Lorazepam 2mg twice daily
  Interventions: Drug: Lorazepam
- D (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD7325 — 4 tablets and 1 capsule taken twice a day for 28 days
  Arms: A
Drug: AZD7325 — 4 tablets and 1 capsule taken twice a day for 28 days
  Arms: B
Drug: Lorazepam — 4 tablets and 1 capsule taken twice a day for 28 days
  Arms: C
Drug: Placebo — 4 tablets and 1 capsule taken twice a day for 28 days
  Arms: D

SUMMARY:
The purpose of this research study is to determine whether AstraZeneca's drug AZD7325 is safe and effective in the treatment of generalized anxiety disorder.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent before any study-related procedures start.
* The patient is previously diagnosed with Generalized Anxiety Disorder.
* The patient has a HADS-A (anxiety) score ≥10 at both screening and randomization.

Exclusion Criteria:

* Patient has a lifetime history of schizophrenia or other psychotic disorders
* Patient has a history of seizures or seizure disorder.
* Patient is pregnant or breast feeding.
* Patient has received electroconvulsive treatment (ECT) in the past.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 369 (Actual)
Dates: Start 2008-12; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark A. Smith, MD, PhD, Study Director — AstraZeneca
Locations (51):
- United States (51):
  - Research Site, Mesa, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, Carson, California
  - Research Site, Escondido, California
  - Research Site, Glendale, California
  - Research Site, Irvine, California
  - Research Site, Redlands, California
  - Research Site, Riverside, California
  - Research Site, Sherman Oaks, California
  - Research Site, Fort Lauderdale, Florida
  - Research Site, Fort Myers, Florida
  - Research Site, Gainsville, Florida
  - Research Site, Hallandale, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Maitland, Florida
  - Research Site, Orlando, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Tampa, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Hoffman Estates, Illinois
  - Research Site, Oak Brook, Illinois
  - Research Site, Schaumburg, Illinois
  - Research Site, Lafayette, Indiana
  - Research Site, Terre Haute, Indiana
  - Research Site, Shreveport, Louisiana
  - Research Site, Glen Burnie, Maryland
  - Research Site, Westminster, Maryland
  - Research Site, Braintree, Massachusetts
  - Research Site, Piscataway, New Jersey
  - Research Site, Cedarhurst, New York
  - Research Site, New York, New York
  - Research Site, Staten Island, New York
  - Research Site, Raleigh, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Willoughby, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Eugene, Oregon
  - Research Site, Salem, Oregon
  - Research Site, Allentown, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Charleston, South Carolina
  - Research Site, Bartlett, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Wichita Falls, Texas
  - Research Site, Richmond, Virginia
  - Research Site, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: International multi-center study, 43 sites recruited between Dec 2008 and May 2009
Pre-assignment Details: Screening for eligibility and wash-out of restriced medications
Groups:
- AZD7325 5 mg: AZD7325 5 mg twice daily (BID)
- AZD7325 15 mg: AZD7325 15 mg twice daily (BID)
- Lorazepam: Lorazepam 2 mg twice daily (BID)
- Placebo: Placebo
Period: Overall Study
Arm/Group | AZD7325 5 mg | AZD7325 15 mg | Lorazepam | Placebo
Started | 93 | 92 | 92 | 92
Completed | 66 | 67 | 78 | 77
Not Completed | 27 | 25 | 14 | 15
Not completed — Adverse Event | 12 | 12 | 5 | 4
Not completed — Protocol Violation | 4 | 5 | 3 | 3
Not completed — Withdrawal by Subject | 5 | 4 | 1 | 4
Not completed — Lost to Follow-up | 4 | 0 | 2 | 1
Not completed — Lack of Efficacy | 0 | 0 | 1 | 2
Not completed — Intake of prohibited medicine | 0 | 0 | 2 | 0
Not completed — All other reasons (not provided) | 2 | 4 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD7325 5 mg | AZD7325 15 mg | Lorazepam | Placebo | Total
Number analyzed (Participants) | 93 | 92 | 92 | 92 | 369
Age, Customized [Number; unit: Participants]
  18-39 years | 46 | 42 | 43 | 44 | 175
  40-65 years | 47 | 50 | 49 | 48 | 194
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 43 | 45 | 45 | 191
  Male | 35 | 49 | 47 | 47 | 178

OUTCOME MEASURES:

1. Primary Outcome: Change in the Hamilton Rating Scale for Anxiety (HAM-A) Total Score
Description: HAM-A total score 0-56 units, 14 questions scored on scale of 0-4 (0= Not present, 4=Very severe) . Higher HAM-A scores indicate higher levels of anxiety Change : score at week 4 minus score at randomization
Time Frame: Baseline to week 4
Measure: Least Squares Mean (Standard Error); unit: Units on scale
Arm/Group | AZD7325 5 mg | AZD7325 15 mg | Lorazepam | Placebo
Number analyzed (Participants) | 89 | 89 | 91 | 90
Units on scale | -10.1 (0.89) [lower limit 0.89] | -10.4 (0.89) [lower limit 0.89] | -10.8 (0.88) [lower limit 0.88] | -9.5 (0.88) [lower limit 0.88]

2. Secondary Outcome: Change in Hospital Anxiety and Depression Scale for Anxiety (HADS-A) Total Score
Description: HADS-A total score 0-21 units, 0 is the best, Higher total scores indicate a higher severity of the mood or anxiety disorder Change : score at week 4 minus score at randomization
Time Frame: Baseline to week 4
Measure: Least Squares Mean (Standard Error); unit: Units on scale
Arm/Group | AZD7325 5 mg | AZD7325 15 mg | Lorazepam | Placebo
Number analyzed (Participants) | 89 | 89 | 91 | 90
Units on scale | -5.0 (0.51) [lower limit 0.51] | -4.9 (0.51) [lower limit 0.51] | -5.0 (0.51) [lower limit 0.51] | -4.5 (0.50) [lower limit 0.50]

3. Secondary Outcome: Change in Psychic Anxiety Factor as Measured by HAM-A Psychic Cluster Score
Description: The HAM-A psychic anxiety cluster score 0-28 units consists of 7 questions scored on scale of 0-4 (0=Not present, 4=Very severe) . Higher scores indicate higher levels of psychic anxiety disorder.
  Change: score at week 4 minus score at randomization
Time Frame: Baseline to week 4
Measure: Least Squares Mean (Standard Error); unit: Units on scale
Arm/Group | AZD7325 5 mg | AZD7325 15 mg | Lorazepam | Placebo
Number analyzed (Participants) | 89 | 89 | 91 | 90
Units on scale | -5.5 (0.51) [lower limit 0.51] | -5.7 (0.51) [lower limit 0.51] | -6.0 (0.51) [lower limit 0.51] | -5.1 (0.51) [lower limit 0.51]

4. Secondary Outcome: Change in Somatic Symptoms as Measured by HAM-A Somatic Cluster Score
Description: The HAM-A Somatic cluster score 0-28 units consists of 7 questions scored on scale of 0-4 (0=Not present, 4=Very severe ) . Higher scores indicate higher levels of psychic anxiety disorder.
Time Frame: Baseline to week 4
Measure: Least Squares Mean (Standard Error); unit: Units on scale
Arm/Group | AZD7325 5 mg | AZD7325 15 mg | Lorazepam | Placebo
Number analyzed (Participants) | 89 | 89 | 91 | 90
Units on scale | -4.5 (0.43) [lower limit 0.43] | -4.7 (0.43) [lower limit 0.43] | -4.9 (0.43) [lower limit 0.43] | -4.3 (0.43) [lower limit 0.43]

5. Secondary Outcome: Change in Quality of Life Enjoyment and Satisfaction Questionnaire Short Form (Q-LES-Q-SF) Percent Maximum Total Score
Description: Q-LES-Q total score is the sum of the first 14 times of Q-LES-Q, and this total score is converted to a % maximum total score by : Q-LES-Q total score /70 x 100%, Larger values indicate a higher perceived quality of life enjoyment and satisfaction.
  Change : percentage at week 4 minus percentage at randomization
Time Frame: Baseline to week 4
Measure: Least Squares Mean (Standard Error); unit: percentage
Arm/Group | AZD7325 5 mg | AZD7325 15 mg | Lorazepam | Placebo
Number analyzed (Participants) | 88 | 89 | 91 | 90
percentage | 7.79 (1.339) [lower limit 1.339] | 9.04 (1.338) [lower limit 1.338] | 7.46 (1.318) | 6.95 (1.317) [lower limit 1.317]

ADVERSE EVENTS:
Arm/Group | AZD7325 5 mg | AZD7325 15 mg | Lorazepam | Placebo
Serious Adverse Events (participants affected / at risk) | 0/93 | 0/92 | 0/92 | 0/92
Other Adverse Events (participants affected / at risk) | 63/93 | 59/92 | 65/92 | 51/92
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AZD7325 5 mg (N=93) | AZD7325 15 mg (N=92) | Lorazepam (N=92) | Placebo (N=92)
Nausea (Gastrointestinal disorders) | 11 | 8 | 7 | 8
Diarrhoea (Gastrointestinal disorders) | 3 | 7 | 5 | 5
Dry Mouth (Gastrointestinal disorders) | 4 | 5 | 6 | 3
Vomiting (Gastrointestinal disorders) | 3 | 1 | 2 | 5
Fatigue (General disorders) | 10 | 2 | 15 | 8
Feeling Abnormal (General disorders) | 5 | 8 | 4 | 3
Feeling Drunk (General disorders) | 5 | 4 | 5 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 5 | 1 | 6
Increased Appetite (Metabolism and nutrition disorders) | 5 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 31 | 27 | 14 | 11
Somnolence (Nervous system disorders) | 18 | 16 | 29 | 11
Headache (Nervous system disorders) | 8 | 8 | 11 | 11
Sedation (Nervous system disorders) | 3 | 6 | 7 | 1
Euphoric Mood (Psychiatric disorders) | 8 | 7 | 4 | 1
Anxiety (Psychiatric disorders) | 5 | 3 | 1 | 1
Mood Altered (Psychiatric disorders) | 5 | 4 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other